

#### PARTICIPANT CONSENT FORM

Music listening for wellbeing in adults with acquired visual impairment who experience anxiety and/or stress and/or depression.

# Main investigator and contact details:

**Nurbanu Somani** (<u>nurbanu.somani@pgr.aru.ac.uk</u>) *Postgraduate researcher, ARU Cambridge* 

Members of the research team:

# **Professor Peter Allen**

Director of Vision and Hearing Research Centre, ARU Cambridge (Principal supervisor)

## **Dr Eldre Beukes**

Senior Lecturer, Vision and Hearing Sciences ARU Cambridge (Supervisor)

## **Dr Alex Street**

Senior Research Fellow, Cambridge institute for Music Therapy Research, ARU Cambridge (Supervisor)

- 1. I confirm I am 18 years of age or older
- 2. I have acquired sight loss (someone who has lost part or all their sight later in life)
- 3. I do not have a hearing impairment that renders I am unable to listen to music and follow a conversation on the telephone.
- 4. I am familiar with using a streaming platform to listen to music online.
- 5. I agree to be contacted after the study is completed, to be invited to participate in a optional one-to-one interview via Zoom or telephone.
- 6. I agree to take part in the above research. I have read the Participant Information Sheet (10/12/21, V1.1) for the study.
- 7. I understand the time involved in completing this study.
- 8. I understand what my role will be in this research, and all my questions have been answered to my satisfaction.
- 9. I agree to be informed and signposted to seek further support if my scores are higher than the normal range.
- 10. I understand words and quotes from my survey or interview responses will be pseudo-anonymised when presenting the findings from this study in the researcher

Nurbanu Somani's thesis, research conferences and publications.

- 11. I understand that I am free to withdraw from the research at any time, without giving a reason.
- 12. I am free to ask any questions at any time before and during the study.
- 13. I understand what information will be collected from me for the study.
- 14. For the purposes of the Data Protection Act (2018), if this project requires me to produce personal data, I have read and understood how Anglia Ruskin University will process it.
- 15. I understand what will happen to the data collected from me for the research.
- 16. I have been told about any disadvantages or risks regarding me taking part.
- 17. I understand that the interviews will be recorded
- 18. I have been provided with a copy of this form and the Participant Information Sheet (10/12/21, V1.1)

Please select here if you agree with the above, or please close the window to exit from this study if you do not agree. (Consent via Qualtrics)